CLINICAL TRIAL: NCT05589519
Title: Rehabilitation of Partial Edentulism Through the Use of Polyetheretherketone (PEEK) Prosthetic 3' Unit Fixed Prosthesis Supported by Dental Implants.
Brief Title: Partial Implant-supported Rehabilitation Using PEEK
Acronym: PEEKPilotSB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Invibio Ltd decided to leave the market and stop PEEK production
Sponsor: Malo Clinic (Other)
Collaborators: Invibio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEEKPilotSB
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Prosthesis Survival
Keywords: prosthesis; dental implants; PEEK
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Partial rehabilitation using PEEK (Experimental): A 3-unit implant-supported fixed prosthesis using PEEK polymer in its composition for the rehabilitation of the partial edentulous.
  Interventions: Device: Partial rehabilitation using PEEK

INTERVENTIONS:
Device: Partial rehabilitation using PEEK — A 3-unit implant-supported fixed prosthesis using PEEK polymer in its composition delivered as definitive prosthesis for partial rehabilitation of edentulous jaws.
  Other Names: PEEK prosthesis

SUMMARY:
The goal of this observational study is to evaluate the outcome of a Poly-ether-ether-ketone - used in partial implant-supported rehabilitations after one year of follow-up. The main question it aims to answer is:

- What is the survival outcome of partial implant-supported prosthesis using Poly-ether-ether-ketone? The participants already rehabilitated with dental implants will receive a definitive 3 unit prosthesis incorporating Poly-ether-ehter-ketone.

DETAILED DESCRIPTION:
Following the previous study on the full-arch rehabilitation of edentulous jaws using hybrid prostheses with polyetheretherketone (PEEK) infrastructure and acrylic resin teeth supported by implants in immediate function inserted through the All-on-4 concept it is necessary to further extend the evaluation to the partial rehabilitation using 3 Unit fixed prostheses supported by dental implants. To test this, the study design to be used will be a single-centre, prospective, observational cohort study to evaluate the short term outcome of fixed prosthetic implant-supported rehabilitations. The sample of this study consists in 10 patients consecutively treated. The cohort will be evaluated at 4 to 8 weeks, 6 months and 12 months after dental loading and annually thereafter as long as the patient is willing, regarding: prosthetic survival including repair and relining, implant survival, marginal bone resorption, incidence of mechanical complications [loosening or fracture of prosthetic components), biological complications (peri-implant infection, suppuration, abscess, fistulae), patient tissue reaction, aesthetic examination including denture staining, colour stability and anatomic form; patients' in-mouth comfort and quality of life using the Oral Health Impact Profile OHIP-14 questionnaire; and assessment of prosthetic preparation (technician satisfaction), laboratory preparation time, clinical operative time and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients rehabilitated with dental implants and a 3 unit Bridge where the molars are missing in one jaw, with at least both canines present;
* Subjects who, in the opinion of the Investigator, are able to understand this clinical study, co-operate with the procedures and are willing to return to the clinic for all the required post-operative follow-ups;
* Subjects who are able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained.

Exclusion Criteria:

* Female Subjects who are pregnant;
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-ups or treatment outcomes;
* Subjects who are currently enrolled in a clinical study;
* Subjects requiring or currently having ongoing orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Survival of the prosthesis | one year
  Evaluation of the survival for the implant-supported prosthesis; nominal (survival,failure)

SECONDARY OUTCOMES:
Survival of the implants | one year
  Evaluation of the survival for implants supporting the PEEK-acrylic resin implant-supported prosthesis; nominal (survival,failure)
Incidence of biological complications | one year
  Peri-implant infection, abscess, fistulae, suppuration, sinus infection, gingival dehiscence; Nominal (no incidence, incidence)
Incidence of mechanical complications | one year
  Loosening or fracture of prosthetic components; Nominal (no incidence, incidence)
Marginal bone resorption | one year
  Measured through periapical radiographs, in mm between the implant shoulder and the most apical portion of implant-bone contact; Scale
Denture staining | one year
  Veneer staining; 0:heavily stained; 10: no stains
Denture colour stability | one year
  Veneer colour stability. Visual analoge scale (0-10 cm); 0: heavily destabilized colour; 10: complete colour stability
Denture anatomic form | one year
  Anatomic form stability. Visual analogue scale (0-10 cm); 0: heavy loss of anatomical shape; 10: complete anatomic stability.
Patient tissue reaction | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
ln mouth comfort | one year
  Patient in mouth comfort. Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Oral Health Impact Profile OHIP-14 | one year
  Oral Health Impact Profile OHIP-14 questionnaire
Laboratory preparation time | one year
  Average laboratory time to produce the finished prosthesis, the active technician time spent in Computer assisted design, Computer assisted manufacture, mill and veneering.
Clinical operative time | one year
  Average operative time to load the final prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Principal Investigator — Director of Research, Development and Education
Locations (1):
- Malo Clinic, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized database containing the study variables
Supporting Information: SAP
Time Frame: Upon study completion and for 8 years.
Access Criteria: Upon solicitation to the Investigators